CLINICAL TRIAL: NCT05260996
Title: Observational Studies About Implementing a Sexual Health Curriculum in Adolescents ( "Big Decisions") of the Canton Riobamba, Chimborazo - Ecuador
Brief Title: Big Decisions - an Evaluation of a Comprehensive Sexual Health Curriculum Pilot in Ecuador During 2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National University of Chimborazo, Riobamba Ecuador (Unknown)
Responsible Party: Principal Investigator, Garrett Kneese, Student, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-18-0979
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Adolescent Sexual Behavior
Keywords: Adolescence; reproductive health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Group (Experimental)
  Interventions: Other: Pilot Group
- Control Group (No Intervention)

INTERVENTIONS:
Other: Pilot Group — 12 Weeks, 1-1 Hour Session Per Week for 10 Total Curriculum Sessions,including 1 Week of Orientation and 1 Week of Debriefing/Program Graduation.
  Arms: Pilot Group

SUMMARY:
The purpose of this study is to assess the efficacy of the "Big Decisions" Adolescent sexual and reproductive health (ASRH) Curriculum via a pilot program with an educational experimental trial design.

ELIGIBILITY:
Inclusion Criteria:

* Student at the Liceo Policial High School in Riobamba, Ecuador(Pilot Site)
* Student at COMIL High school in Riobamba(Control Site)
* Student of 9th or 10th grade.

Exclusion Criteria:

* Not a current student at the Liceo Policial High School in Riobamba, Ecuador(Pilot Site)
* Not a current student at COMIL high school in Riobamba.(Control Site)
* Not a student of 9th or 10th grade.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Qualitative perceptions surrounding self-efficacy as assessed by the General Self-Efficacy Scale. | Baseline
Qualitative perceptions surrounding self-efficacy as assessed by the General Self-Efficacy Scale. | week 12
Qualitative perceptions surrounding gender as assessed by the Gender Equitable Men (GEM) Scale. | Baseline
Qualitative perceptions surrounding gender as assessed by the Gender Equitable Men (GEM) Scale. | week 12
Qualitative perceptions surrounding gender as assessed by the Attitudes Toward Women Scale (AWSA) Scale. | Baseline
Qualitative perceptions surrounding gender as assessed by the Attitudes Toward Women Scale (AWSA) Scale. | week 12
Qualitative perceptions surrounding relational norms as assessed by the Sexual Relationship Power Scale (SRPS) | Baseline
Qualitative perceptions surrounding relational norms as assessed by the Sexual Relationship Power Scale (SRPS). | week 12
Qualitative perceptions surrounding reproductive health knowledge as assessed by the Knowledge, Attitudes, and Practices (Sexual) (KAPS) survey. | Baseline
Qualitative perceptions surrounding reproductive health knowledge as assessed by the Knowledge, Attitudes, and Practices (Sexual) (KAPS) survey. | week 12
Qualitative perceptions surrounding risk behaviors surrounding reproductive health as assessed by the Youth Risk Behavior Surveillance System (YRBSS) survey. | Baseline
Qualitative perceptions surrounding risk behaviors surrounding reproductive health as assessed by the Youth Risk Behavior Surveillance System (YRBSS) survey. | week 12
Percentage of Surveys with 100% Completion of All Questions. | Baseline
  To calculate this percentage, the number of surveys with 100% completion of all questions will be divided by the number of surveys administered.
Percentage of Surveys with 100% Completion of All Questions. | week 12
  To calculate this percentage, the number of surveys with 100% completion of all questions will be divided by the number of surveys administered.
Percentage of Surveys with 100% Completion of All Questions. | week 16
  To calculate this percentage, the number of surveys with 100% completion of all questions will be divided by the number of surveys administered.
Percentage of Surveys with 100% Completion of All Questions. | week 24
  To calculate this percentage, the number of surveys with 100% completion of all questions will be divided by the number of surveys administered.
Number of students who abstain from participating in surveys | week 12
Number of students who abstain from participating in surveys | week 16
Number of students who abstain from participating in surveys | week 24
Number of students who participate in surveys | week 12
Number of students who participate in surveys | week 16
Number of students who participate in surveys | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Kneese, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No